CLINICAL TRIAL: NCT00319293
Title: Efficacy of Metformin in Lean Women With Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 160350-2
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Insulin resistance is an important feature of the polycystic ovary syndrome,and patiens are successfully treated with the insulin sensitizing agent metformin. The insulin resistance of lean patients with the syndrome is debated. In this study, we will study the change in insulin resistance, metabolic and hormonal factors after 3 months of metformin treatment in lean PCOS women.

ELIGIBILITY:
Inclusion Criteria:

* PCOS (Rotterdam criteria)
* BMI < 27
* No medication for 3 months

Exclusion Criteria:

* Pregnancy
* Lactation
* Other endocrinologic disease

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20

PRIMARY OUTCOMES:
Insulin resistance
Hormonal factors
Metabolic factors

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta Trolle, MD, Principal Investigator — Skejby University Hospital